CLINICAL TRIAL: NCT00698672
Title: A Prospective Randomized RSA-Study of Cemented Hip Prostheses With Five Different Articulations
Brief Title: RSA-Study of Cemented Hip Prostheses With Five Different Articulations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10642(NSD); 197.03(REK) (Other: Regional Etisk Komite)
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Arthritis
Keywords: RSA
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- 2 (Active Comparator): articulation Spectron EF CoCr/ Reflection All-Poly Eto-sterilized
  Interventions: Device: Spectron Reflection CoCr
- 3 (Active Comparator): articulation Spectron Ef CoCr/ Reflection All-Poly XLPE
  Interventions: Device: Spectron XLPE CoCr
- 4 (Active Comparator): articulation Spectron EF Oxinium/ Reflection All-Poly Eto-sterilized
  Interventions: Device: Spectron Reflection Oxinium
- 5 (Active Comparator): articulation Spectron EF Oxinium/ Reflection XLPE
  Interventions: Device: Spectron XLPE CoCR
- 1 (Active Comparator): articulation Charnley/ Ogee
  Interventions: Device: charnley OGEE

INTERVENTIONS:
Device: charnley OGEE — charnley OGEE
  Arms: 1
Device: Spectron Reflection CoCr — Spectron Reflection CoCr
  Arms: 2
Device: Spectron XLPE CoCr — Spectron XLPE CoCr
  Arms: 3
Device: Spectron Reflection Oxinium — Spectron Reflection Oxinium
  Arms: 4
Device: Spectron XLPE CoCR — Spectron XLPE CoCR
  Arms: 5

SUMMARY:
The purpose of this study is to compare wear and migration of the following hip prostheses:

1. Charnley monoblock 22.2mm caput and OGEE polyethylene acetabular component
2. Spectron EF stem with Reflection polyethylene cup and 28 mm CoCr caput
3. Spectron EF stem with XLPE cup and 28 mm CoCr caput
4. Spectron EF stem with Reflection polyethylene cup and 28 mm Oxinium caput
5. Spectron EF stem with XLPE cup and 28 mm Oxinium caput

DETAILED DESCRIPTION:
Detailed description in:

Wear and migration of highly cross-linked and conventional cemented polyethylene cups with cobalt chrome or Oxinium femoral heads: a randomized radiostereometric study of 150 patients.

Kadar T, Hallan G, Aamodt A, Indrekvam K, Badawy M, Skredderstuen A, Havelin LI, Stokke T, Haugan K, Espehaug B, Furnes O.

J Orthop Res. 2011 Aug;29(8):1222-9. doi: 10.1002/jor.21389

ELIGIBILITY:
Inclusion Criteria:

* arthritis
* dysplasia

Exclusion Criteria:

* obesitas
* charcots
* paget
* malignancy

Ages: 59 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-11; Primary Completion 2007-06 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
wear | 2 years

SECONDARY OUTCOMES:
migration | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kadar, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
Not planned

REFERENCES:
- [Derived] Johannessen HG, Hallan G, Kadar T, Lie SA, Lygre SHL, Fenstad AM, Haugan K, Hol PJ, Badawy M, Jonsson B, Indrekvam K, Aamodt A, Furnes O. Early cup migration and wear as predictors for later aseptic loosening: a secondary evaluation of a randomized controlled RSA trial on cemented hip arthroplasties with 18-year follow-up. Acta Orthop. 2025 Aug 15;96:618-624. doi: 10.2340/17453674.2025.44328. PMID 40814981